CLINICAL TRIAL: NCT04936295
Title: A Phase II Study of the Efficacy and Tolerability of Fulvestrant Plus Anlotinib in HR(+)/HER2(-) Metastatic Breast Cancer Patients With FGFR Mutation
Brief Title: Fulvestrant Plus Anlotinib in HR(+)/HER2(-) Metastatic Breast Cancer With FGFR Mutation
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, Xu fei, Associate Chief Physician, Sun Yat-sen University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SYSU005
Record Dates: First submitted 2021-06-16; First posted 2021-06-23 (Actual); Last update posted 2021-06-23 (Actual); Status verified 2021-06

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Fulvestrant; anlotinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Fulvestrant plus Anlotinib (Experimental): Each participant receives fulvestrant combined with anlotinib.
  Interventions: Drug: Fulvestrant plus Anlotinib

INTERVENTIONS:
Drug: Fulvestrant plus Anlotinib — Each patient receives Fulvestrant (500mg delivered by intramuscular injection every 4 weeks) plus Anlotinib(20mg taken orally for 14 days and stop for 7 days in one cycle)

SUMMARY:
Previous studies have shown that the FGF signaling pathway is closely related to endocrine therapy resistance in breast cancer, but there is not sufficient evidence for the combination of endocrine therapy and FGFR inhibitors. Anlotinib is a highly effective VEGFRs, FGFRs, PDGFRs multi-target tyrosine kinase inhibitor. Therefore, we conducted this single-arm, single-center phase II clinical study to evaluate the efficacy and the safety of anlotinib combined with fulvestrant in patients with metastatic HR+/HER2- breast cancer patients with FGFR mutation and resistance to aromatase inhibitor therapy, to provide new treatment options for these patients.

DETAILED DESCRIPTION:
Endocrine therapy resistance is an unsolved problem in the treatment of HR+/HER2- metastatic breast cancer. Previous studies have shown that the FGF signaling pathway is closely related to endocrine therapy resistance in breast cancer, but there is not sufficient evidence for the combination of endocrine therapy and FGFR inhibitors. Anlotinib is a highly effective VEGFRs, FGFRs, PDGFRs multi-target tyrosine kinase inhibitor, which can effectively block the migration and proliferation of endothelial cells and reduce tumor microvessel density. The drug inhibits VEGFRs, FGFRs, PDGFRs to exert anti-angiogenesis effects and to achieve anti-tumor effects. Therefore, we conducted this single-arm, single-center phase II clinical study to evaluate the efficacy and the safety of anlotinib combined with fulvestrant in patients with metastatic HR-positive and HER2-negative breast cancer patients with FGFR mutation and resistance to aromatase inhibitor therapy, to provide new treatment options for these patients.

ELIGIBILITY:
Inclusion Criteria:

1. Voluntarily sign the informed consent form;
2. 18-75 years old;
3. Women in any menstrual state, premenopausal or perimenopausal patients need to receive luteinizing hormone releasing hormone(LHRH) analogue;
4. Eastern Cooperative Oncology Group (ECOG) score [0-1] points;
5. The expected survival period is ≥12 weeks;
6. The diagnosis of invasive carcinoma by histology or cytology; Estrogen receptor (ER) positive (defined as >1% nuclear ER staining); HER2 negative (defined as IHC 0 or 1+, or HER2(2+) with HER2 FISH detection no amplification);
7. Inoperable or recurrent/metastatic breast cancer patients with aromatase inhibitor treatment failure;
8. In the state of disease progression before enrollment;
9. There are FGFR mutations, which meets any of the following: ①Immunohistochemical method: any subtype of FGFR1/2/3/4 is positive; ② Gene detection results of tissue/blood sample shows that any subtype of FGFR1/2/3/4 has functional variation such as amplification, activating mutation or fusion;
10. Measurable disease according to RECIST version 1.1 or only bone metastasis;
11. Adequate hematological, hepatic function;
12. Doppler ultrasound: left ventricular ejection fraction (LVEF) ≥50%.

Exclusion Criteria:

1. Have used Fulvestrant or its analogues;
2. History of other primary malignancy;
3. Allergic to the ingredients of Anlotinib Hydrochloride Capsules;
4. Previously received targeted drug therapy for FGFR;
5. Received chemotherapy within 4 weeks before enrollment;
6. Received endocrine therapy within 2 weeks before enrollment;
7. Patients with currently symptomatic brain or meningeal metastasis;
8. Concomitant diseases/conditions that is not controllable, and any other major illness that, in the investigator's judgment, will substantially increase the risk associated with the patient's participation in this study;
9. Patients who cannot accept drugs orally;
10. Any other situation that the investigator judges cannot be enrolled in the study.

Ages: 18 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 61 (Estimated)
Dates: Start 2021-06-16 (Estimated); Primary Completion 2023-06-01 (Estimated); Study Completion 2025-06-01 (Estimated)

PRIMARY OUTCOMES:
Clinical benefit rate (CBR) | 24 weeks
  Response and progression will be evaluated using RECIST 1.1. Evaluation will occur every 3 months till progression or termination of the study. CBR is defined as ratio of participants who have stable disease for over 24 weeks.

SECONDARY OUTCOMES:
Progression free survival (PFS) | 1 year
  Time from the date of treatment to the date of tumor progression
Objective response rate (ORR) | 1 year
  The proportion of best overall response of either complete or partial response.
Overall survival (OS) | 3 years
  Time from the date of treatment to the date of death.
Number of Participants with Adverse Events | 1 year
  Number of participants with adverse events related to the treatment.
The quality of life | 1 year
  Using EORTC (European Organization for Research and Treatment of Cancer) QLQ-BR23 scale. The minimum and maximum values are 0 and 100, respectively. Higher scores mean better outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Fei Xu, MD, Principal Investigator — Sun Yat-sen University
Locations (1):
- Sun Yat-sen University Cancer Center, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No